CLINICAL TRIAL: NCT06184269
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 4-period, Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1017-1" and Co-administration of "BR1017-1A" and "BR1017-1B" in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1017-1" and Co-administration of "BR1017-1A" and "BR1017-1B"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FAEC-CT-102
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Essential Hypertension; Primary Hypercholesterolemia
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1017-1A+BR1017-1B (Active Comparator)
  Interventions: Drug: BR1017-1A; Drug: BR1017-1B
- BR1017-1 (Experimental)
  Interventions: Drug: BR1017-1

INTERVENTIONS:
Drug: BR1017-1 — One tablet administered alone
  Arms: BR1017-1
Drug: BR1017-1A — One tablet administered alone
  Arms: BR1017-1A+BR1017-1B
Drug: BR1017-1B — One tablet administered alone
  Arms: BR1017-1A+BR1017-1B

SUMMARY:
The objective of this clinical study is to evaluate the pharmacokinetics and the safety after administration of "BR1017-1" and co-administration of "BR1017-1A" and "BR1017-1B" in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who weigh 50 kg or more and have body mass index (BMI) within the range of 18.0 to 30.0kg/m² at screening visit.
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken drugs concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months prior to the first administration date.(However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal surgery or gastrointestinal diseases that may affect the absorption of drugs. (Except for simple appendectomy, hernia surgery)
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or its products) that may affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours prior to the first day of administration.
* In the case of a female subject, those suspected pregnancy, pregnant woman, lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0-72 hours after administration
  Area under the concentration-time curve from time zero to time τ
Cmax | 0-72 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No